CLINICAL TRIAL: NCT02023463
Title: Phase Ib Trial of Enzalutamide in Combination With Radiation Therapy and LHRH Agonist Therapy in the Management of Intermediate and High-Risk Prostate Cancer
Brief Title: Enzalutamide, Radiation Therapy and Hormone Therapy in Treating Patients With Intermediate or High-Risk Prostate Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Collaborators: Astellas Pharma Inc (Industry); Medivation, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13P.461; 2013-027 (Other: CCRRC); JT 2970 (Other: JeffTrial Number)
Record Dates: First submitted 2013-12-23; First posted 2013-12-30 (Estimated); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Adenocarcinoma of the Prostate; Recurrent Prostate Cancer; Stage IIB Prostate Cancer; Stage III Prostate Cancer; Stage IV Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — enzalutamide; Goserelin; Leuprolide; Radiotherapy; Radiation; Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (enzalutamide, radiation therapy, hormone therapy) (Experimental): Patients receive enzalutamide PO QD for 6 months. Beginning 2 weeks after start of enzalutamide, patients receive LHRH agonist therapy with goserelin acetate SC or leuprolide acetate IM or SC for 6 months (intermediate risk patients) or 24 months (high risk patients) post-radiation therapy. Beginning 8 weeks after the start of LHRH therapy, patients undergo either IMRT or VMAT daily five days a week for 8 weeks.
  Interventions: Drug: Enzalutamide; Drug: Goserelin acetate; Drug: Leuprolide acetate; Radiation: Radiation therapy

INTERVENTIONS:
Drug: Enzalutamide — Given PO
  Other Names: Xtandi; MDV3100
Drug: Goserelin acetate — Given SC
  Other Names: Goserelin; Zoladex
Drug: Leuprolide acetate — Given IM or SC
  Other Names: Leuprorelin; Leuprolide
Radiation: Radiation therapy — Undergo image-guided radiation therapy
  Other Names: irradiation; radiotherapy; therapy; radiation

SUMMARY:
This phase I trial studies the side effects and best way to give enzalutamide, radiation therapy, and hormone therapy in treating patients with intermediate or high-risk prostate cancer. Androgens can cause the growth of prostate cancer cells. Antihormone therapy, such as enzalutamide, may lessen the amount of androgens made by the body. Radiation therapy uses high energy x rays to kill tumor cells. Giving enzalutamide, radiation therapy, and hormone therapy may be an effective treatment for prostate cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

1) To assess the safety of the combination of neoadjuvant and concurrent enzalutamide with an luteinizing-hormone-releasing hormone (LHRH) agonist and radiation therapy.

SECONDARY OBJECTIVES:

1. To determine the efficacy of the combination of enzalutamide with an LHRH agonist and radiation therapy using prostate specific antigen (PSA) kinetics.
2. To determine the efficacy of the combination of enzalutamide with an LHRH agonist and radiation therapy using PSA nadir.
3. To describe patient-reported outcomes including: Expanded Prostate Cancer Index Composite (EPIC), American Urological Association (AUA) Symptom Index, PROstate magnetic resonance (MR) Imaging Study (PROMIS) Fatigue Scale.

OUTLINE:

Patients receive enzalutamide orally (PO) once daily (QD) for 6 months. Beginning 2 weeks after start of enzalutamide, patients receive LHRH agonist therapy with goserelin acetate subcutaneously (SC) or leuprolide acetate intramuscularly (IM) or SC for 6 months (intermediate risk patients) or 24 months (high risk patients) post-radiation therapy. Beginning 8 weeks after the start of LHRH agonist therapy, patients undergo either intensity modulated radiation therapy (IMRT) or volumetric arc therapy (VMAT) daily five days a week for 8 weeks.

After completion of study treatment, patients are followed up every 3 months for 2 years, every 6 months for 2 years, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

1. Prostate adenocarcinoma without distant metastatic disease with either Gleason score ≥ 7, PSA ≥ 10 ng/ml, or T2b or greater disease
2. Age > 18
3. Performance Status: ECOG 0-1
4. Hematologic (minimal values):

   * Absolute neutrophil count > 1,500/mm3
   * Hemoglobin > 8.0 g/dl
   * Platelet count > 100,000/mm3
5. Hepatic function

   * Total bilirubin < Upper limit of normal (ULN)(except for Gilbert's disease)
   * AST (SGOT) < 1.5 x ULN
   * ALT (SGPT) < 1.5 x ULN
6. Creatinine < 1.5 x ULN
7. Men of childbearing potential must be willing to consent to using effective contraception while on treatment and for at least 3 months thereafter.

Exclusion Criteria:

1. Patients with a history of seizure, underlying brain injury with loss of consciousness, transient ischemic attack within the past 12 months, cerebral vascular accident, brain metastases, brain arteriovenous malformation or the use of concomitant medications that may lower the seizure threshold
2. History of urological surgery or procedures predisposing to GU complications after radiation (will be determined by radiation oncologist)
3. History of diverticulitis, rectal bleeding or other lower GI diseases predisposing to GI complications after radiation (will be determined by radiation oncologist)
4. History of prior chemotherapy or pelvic irradiation,
5. History of prior invasive malignant cancer(s) within the last 5 years except adequately treated or controlled basal cell or squamous cell carcinoma of the skin.
6. Documented distant metastatic disease. NOTE: pelvic lymphadenopathy is NOT excluded.
7. Prior radical prostatectomy or cryosurgery for prostate cancer or bilateral orchiectomy.
8. No experimental medications within 30 days of study entry
9. Patients currently taking the following medications:

   * CYP2C8 inhibitors (e.g. Gemfibrozil)
   * CYP2C8 inducers (e.g. rifampin)
   * CYP3A4 inhibitors (itraconazole)
   * CYP3A4 inducers (e.g., carbamazepine, phenobarbital, phenytoin, rifabutin, rifampin, rifapentine)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2014-04-02 (Actual); Primary Completion 2017-07-10 (Actual); Study Completion 2040-01-01 (Estimated)

PRIMARY OUTCOMES:
Acute toxicities, monitored using the National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0 criteria | Up to 1 month post completion of enzalutamide
  An exact 2-sided binomial 90% confidence interval will be computed and reported. Toxicity will be monitored and if there is greater than 10% incidence of grade 3 or higher gastrointestinal (GI)/genitourinary (GU)/fatigue lasting more than 7 days despite optimal treatment, the trial will be re-evaluated.

SECONDARY OUTCOMES:
Change in PSA levels | Baseline up to 6 months
  Evaluated using linear mixed models. Mixed models will make use of all available data, and can estimate individual levels of change.
Quality of life (QoL), measured using the EPIC, AUA symptom index, and the PROMIS Fatigue Scale | Baseline up to 1 year
  QoL measures will also be assessed via linear mixed models, as an exploratory evaluation of potential clinical correlates, such as age, race, stage, Gleason score, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Den, MD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States

REFERENCES:
- See also: Thomas Jefferson University Hospitals — http://www.JeffersonHospital.org